CLINICAL TRIAL: NCT05900193
Title: Activation and Inhibition of the Sweet Taste Receptor T1R2-T1R3 Differentially Affect Glucose Tolerance in Humans
Brief Title: Sucralose and Lactisole Additions to OGTT in Humans
Acronym: SLOGTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Paul Breslin, PhD, Professor, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 16-105mc
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Neat OGTT; OGTT With Added Sucralose; OGTT With Added Lactisole

STUDY DESIGN:
Intervention Model Description: Participants were given oral glucose tolerance tests alone or with lactisole or sucralose in admixture with the glucose. All controls were within subjects in counterbalanced crossover design.
Who Masked: Participant, Outcomes Assessor
Masking Description: Plasma levels of glucose and hormones were analyzed without knowledge of condition participant was tested. Participants did not know their condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants receiving oral glucose tolerane tests with TAS1R agonists (Experimental): Participants received a standard oral glucose tolerance test alone and with the addition of the TAS1R2/3 agonist sucralose in admixture
  Interventions: Dietary Supplement: TAS1R2/3 agonist or antagoinst admixture to oral glucose tolerance test
- Participants receiving oral glucose tolerane tests with TAS1R antagonists (Experimental): Participants received a standard oral glucose tolerance test alone and with the addition of the the TAS1R2/3 antagonist lactisole in admixture
  Interventions: Dietary Supplement: TAS1R2/3 agonist or antagoinst admixture to oral glucose tolerance test

INTERVENTIONS:
Dietary Supplement: TAS1R2/3 agonist or antagoinst admixture to oral glucose tolerance test — Participants drank a glucose beverage for an oral glucose tolerance test along or with admixture with the TAS1R2/3 agonist sucralose or the TAS1R2/3 antagonist lactisole.

SUMMARY:
In the present study, our objective was to determine whether T1R2-T1R3 influences glucose metabolism bidirectionally via hyperactivation with sucralose and inhibition with sodium lactisole in mixture with glucose loads during tolerance tests in humans. In 12 healthy participants we conducted oral glucose tolerance tests (OGTTs) of 75 g glucose with and without the addition of the T1R2-T1R3 agonist, sucralose (5 mM). We also conducted OGTTs in 10 healthy participants with and without the addition of a T1R2-T1R3 antagonist, sodium lactisole (2 mM). Plasma glucose, insulin, and glucagon were measured before, during, and after OGTTs up to 120 minutes post-prandially. We also assessed individual participants' sweet taste responses to sucralose, their sensitivities to sweetness inhibition by lactisole, and their BMIs.

DETAILED DESCRIPTION:
The sweet taste receptor, T1R2-T1R3, is expressed in taste bud cells, where it conveys sweetness, and also in intestinal enteroendocrine cells, where it may facilitate glucose absorption and assimilation. There is evidence in mice through genetic knockout studies that T1r2-T1r3 is involved in endocrine and enteroendocrine responses to glucose loads. Yet, our understanding of the impact of T1R2-T1R3 on human glucose metabolism is less clear. In the present study, our objective was to determine whether T1R2-T1R3 influences glucose metabolism bidirectionally via hyperactivation with sucralose and inhibition with sodium lactisole in mixture with glucose loads during tolerance tests in humans. In 12 healthy participants we conducted oral glucose tolerance tests (OGTTs) of 75 g glucose with and without the addition of the T1R2-T1R3 agonist, sucralose (5 mM). We also conducted OGTTs in 10 healthy participants with and without the addition of a T1R2-T1R3 antagonist, sodium lactisole (2 mM). Plasma glucose, insulin, and glucagon were measured before, during, and after OGTTs up to 120 minutes post-prandially. We also assessed individual participants' sweet taste responses to sucralose, their sensitivities to sweetness inhibition by lactisole, and their BMIs. The addition of sucralose to glucose elevated plasma insulin responses to the OGTT. Sucralose-sensitive participants, those who rated sucralose as sweetest, had a more pronounced elevation in peak plasma insulin to sucralose + glucose with early increases in plasma glucose and insulin area-under-the-curve (AUC) within the first 15 minutes. In lactisole-sensitive participants, whose sweetness was suppressed by low levels of lactisole, the addition of lactisole to glucose in the OGTT decreased plasma glucose AUC. Participants with higher BMI (>24 kg/m2) tended to be hyper-responsive to added sucralose, nearly doubling their peak levels of insulin to the sucralose + glucose OGTT . Manipulation of the T1R2-T1R3 receptor with a non-caloric agonist and an antagonist demonstrates that T1R2-T1R3 helps regulate glucose handling and metabolism in humans. Importantly, participants with BMI > 24 kg/m2 tended to rate sucralose as sweeter and showed exaggerated insulin increases when it was added to their OGTT.

ELIGIBILITY:
Inclusion Criteria:

* Non-diabetic
* No metabolic disease
* Should not have exercised in past 24 hours.
* Should have undergone overnight fast.
* BMI <30 kg/m2

Exclusion Criteria:

* Participants who reported consuming more than one serving of artificially sweetened beverages or snacks per day were excluded.
* Participants with diseases (e.g. metabolic syndrome and diabetes) and medications that may affect taste, digestion and absorption (e.g. anti-hypertensives, antibiotics, insulin, metformin, SGLT2 Inhibitors, sulfonylureas) were also excluded.
* Participants with BMI>30 kg/m2 were excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-07-17 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Plasma Glucose | 90 minutes
  Repeated plasma blood draws during OGTT will determine plasma glucose
Plasma Insulin | 90 minutes
  Repeated plasma blood draws during OGTT will determine plasma insulin
Plasma glucagon | 90 minutes
  Repeated plasma blood draws during OGTT will determine plasma glucagon

SECONDARY OUTCOMES:
Taste responsivity to sucralose | 30 minutes
  How sweet sucralose tastes to participants is reported
Taste inhibition by lactisole | 30 minutes
  How effectively lactisole inhibits sweet taste for individual participants is assessed
Body-mass Index | 15 minutes
  Individual participant BMI was calculated

CONTACTS AND LOCATIONS:
Overall Officials: Paul Breslin, PhD, Principal Investigator — Rutgers, The State University of NJ
Locations (1):
- Rutgers, Department of Nutritional Sciences, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Journals require de-identified data be made available to others.
Supporting Information: Study Protocol, SAP
Time Frame: Available upon request
Access Criteria: Contact the PI at breslin@monell.org